CLINICAL TRIAL: NCT03012373
Title: Efficacy of Acupuncture as an Adjunct to Methadone Treatment Services for Heroin Addicts
Acronym: AAMTH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Lu-Tung Christian Hospital (Other)
Responsible Party: Principal Investigator, Wen-Chen Ouyang, Superintendent, Lu-Tung Christian Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LuTungCH-1
Record Dates: First submitted 2016-10-29; First posted 2017-01-06 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Opiate Withdrawal Syndrome
Keywords: methadone; heroin; acupuncture
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ear acupressure & Electroacupuncture (A) (Experimental): Electroacupuncture plus Ear acupressure or Ear acupressure alone for four weeks followed by an one week wash-out period. Then with crossover to the othe.
  Interventions: Procedure: Ear acupressure alone; Procedure: Electroacupuncture plus ear acupressure
- Ear acupressure & Electroacupuncture (B) (Experimental): Electroacupuncture plus Ear acupressure or Ear acupressure alone for four weeks followed by an one week wash-out period. Then with crossover to the othe.
  Interventions: Procedure: Ear acupressure alone; Procedure: Electroacupuncture plus ear acupressure

INTERVENTIONS:
Procedure: Ear acupressure alone — The magnet pellets were placed with adhesive tape at shenmen point of both ears and were pressed 5 times every 5 minutes for 15 minutes then were attached until next treatment and change now one. The patients received this treatment 2 times a week for 4 weeks.
  Other Names: Auricular acupressure
Procedure: Electroacupuncture plus ear acupressure — Acupuncture included Hegu (LI 4) and Zusanli (ST 36) on both hands and legs with electrical stimulation was conducted. The frequency of electrical stimulation was 5 Hz and wave form was adjustable. The intensities of the stimulation were increased in 1 mA increments to maximal tolerable intensity. At the same time, The magnet pellets were placed with adhesive tape at shenmen point of both ears and were pressed 5 times every 5 minutes for 15 minutes. After 15 minutes treatment, acupuncture needles were removed and magnet pellets were attached until next treatment and change now one. The patients received this treatment 2 times a week for 4 weeks.
  Other Names: Electric acupuncture

SUMMARY:
This is an open-label, randomized, 2-sequence, cross-over study evaluating the difference of efficacy between ear acupressure alone and ear acupressure plus electroacupuncture therapy both combined with methadone treatment services for heroin addicts.

DETAILED DESCRIPTION:
Methadone substitution therapy has been the treatment of first choice for opiate dependence, but patient on Methadone substitution therapy report a wide side effects, and relapse rate is up to two third of methadone treatment patients between one to two years. Therefore, adjuvant therapeutic interventions for heroin addiction patients are needed. Since 1996, the World Health Organization (WHO) has classified acupuncture treatment indications, including drug abuse. The purpose of this study is to compare the difference of efficacy between ear acupressure alone and ear acupressure plus electrical acupuncture therapy both combined with standard methadone maintenance therapy to the heroin addicts.

Patients who receive methadone were randomly assigned to sequence A and B. Sequence A(n=20) receive ear Acupressure combined with electroacupuncture for four weeks, followed by one week wash-out period. Then ear acupressure alone for another four weeks.

Sequence B(n=20) receive EAR acupressure alone for four weeks first, and followed by one week wash-out period, then ear acupressure combined with electroacupuncture for another four weeks. Measures of methadone dosage and using the craving visual analog scale (VAS) to assess the craving severity for 8 weeks. Using the Short Form Health Survey (SF-36) and the Pittsburgh Sleep Quality Index (PSQI) to assess improvement of life quality and sleep quality. Using Beck anxiety and Depression inventory to evaluate emotional problems. Urine opiate screenings are provided after 4 weeks , 8 weeks treatment and 1 month after end of treatment, to screen opiate reuse.

The study hypothesis was acupuncture had more clinical efficacy than ear acupressure upon craving severity, life quality, mood stability ,reduced methadone dosage and sleep quality when provided as an adjunct to a standard methadone maintenance treatment.

ELIGIBILITY:
Inclusion Criteria:

Fulfilled Diagnostic and Statistical Manual of Mental Disorders, 5th Edition criteria for Opioid Use Disorder and had been received methadone maintenance treatment for more then one month.

Exclusion Criteria:

1. had taking acupuncture treatment in past 30 days
2. had severe adverse effects or events history from receiving acupuncture treatment
3. had any serious physical illness
4. had a significant risk of suicide
5. ear infection
6. were pregnant or or a woman plan to pregnant
7. had bleeding disorders or were taking anticoagulant drugs
8. had epilepsy, cerebral vascular disease and brain injured history.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-03-30 (Estimated); Study Completion 2018-05-30 (Estimated)

PRIMARY OUTCOMES:
Assessed the change of opioid craving | Four weeks after first phase treatment/ one weeks after washout period/ four weeks after second phase treatment
  opioid craving scores on the Visual Analog Scale

SECONDARY OUTCOMES:
Assessed the change of life quality | Four weeks after first phase treatment/ one weeks after washout period/ four weeks after second phase treatment
  Life quality was assessed using the Taiwanese version of Short Form 36 (SF-36)
Assessed the change of emotion problem | Four weeks after first phase treatment/ one weeks after washout period/ four weeks after second phase treatment
  Emotion problems was evaluated by Beck anxiety and Depression inventory
Opiate usage | Four weeks after first phase treatment/ one weeks after washout period/ four weeks after second phase treatment
  Use urine test to detect opiate use
Assessed the change of sleep quality | Four weeks after first phase treatment/ one weeks after washout period/ four weeks after second phase treatment
  Sleep quality was assessed using the Chinese version of the Pittsburgh Sleep Quality Index (CPSQI)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chen Ouyang, Ph.D., Principal Investigator — Lu-Tung Christian Hospital
Locations (1):
- Lu-Tung Christian Hospital, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chan YY, Lo WY, Li TC, Shen LJ, Yang SN, Chen YH, Lin JG. Clinical efficacy of acupuncture as an adjunct to methadone treatment services for heroin addicts: a randomized controlled trial. Am J Chin Med. 2014;42(3):569-86. doi: 10.1142/S0192415X14500372. PMID 24871652
- [Background] Lin JG, Chan YY, Chen YH. Acupuncture for the treatment of opiate addiction. Evid Based Complement Alternat Med. 2012;2012:739045. doi: 10.1155/2012/739045. Epub 2012 Feb 22. PMID 22474521
- [Background] Boyuan Z, Yang C, Ke C, Xueyong S, Sheng L. Efficacy of acupuncture for psychological symptoms associated with opioid addiction: a systematic review and meta-analysis. Evid Based Complement Alternat Med. 2014;2014:313549. doi: 10.1155/2014/313549. Epub 2014 Nov 4. PMID 25530779